CLINICAL TRIAL: NCT04025710
Title: BIO|MASTER.BIOMONITOR III
Brief Title: Master Study of the BIOMONITOR III and Incision and Insertion Tool (FIT OneStep)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: BA109
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Results first posted 2024-01-11 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2022-11

CONDITIONS: Tachyarrhythmia; Atrial Fibrillation (AF); Syncope; Cryptogenic Stroke
MeSH Terms: conditions — Tachycardia; Atrial Fibrillation; Syncope; Ischemic Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients (Other)
  Interventions: Device: BIOMONITOR III and BIOMONITOR IIIm

INTERVENTIONS:
Device: BIOMONITOR III and BIOMONITOR IIIm — * Insertion of BIOMONITOR III or BIOMONITOR IIIm
  * three scheduled in-office follow-ups
  * 48-hour Holter ECG

SUMMARY:
This study is a post-market clinical follow-up (PMCF) study to identify and evaluate residual risks associated with the use of the BIOMONITOR III and BIOMONITOR IIIm that are discovered or remain even after risk analysis, risk mitigation and successful conformity assessment. Furthermore, this study will also provide additional data as required by regulatory authorities outside of the CE-region.

ELIGIBILITY:
Inclusion Criteria:

* Patient is at high risk of developing a clinically important cardiac arrhythmia; or
* Patient is undergoing investigation for symptoms such as palpitations, pre- syncope or syncope, that are suggestive of an underlying cardiac arrhythmia; or
* Patient is undergoing investigation for the detection of atrial fibrillation following cryptogenic stroke; or
* Patient is planned for AF ablative procedure or has already undergone an AF ablative procedure.
* Patient is able to understand the nature of the study and able to provide written informed consent.
* Patient is willing and able to perform all follow-up visits at the investigational site.
* Patient is willing and able to use the CardioMessenger and accepts the BIOTRONIK Home Monitoring concept.

Exclusion Criteria:

* Patient is implanted with an ICD or pacemaker.
* Patient is pregnant or breast-feeding.
* Patient is less than 18 years old.
* Patient's life-expectancy is less than 12 months.
* Patient is participating in another interventional clinical investigation.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-04-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Deneke, Prof. Dr., Principal Investigator — RHÖN-KLINIKUM Campus Bad Neustadt, Germany
Locations (27):
- Australia (6):
  - GenesisCare Wesley, Auchenflower
  - GenesisCare Bundaberg, Bundaberg
  - GenesisCare Doncaster, Doncaster East
  - Canberra Heart Rhythm Clinic, Garran
  - Prince of Wales Hospital, Randwick
  - Princess Alexandra Hospital, Woolloongabba
- Austria (3):
  - Kepler Universitätsklinikum, Linz
  - Allgemeines Krankenhaus der Stadt Wien (AKH), Vienna
  - Klinikum Wels-Grieskirchen, Wels
- Regionshospitalet Viborg, Viborg, Denmark
- Germany (11):
  - RHÖN-KLINIKUM Campus Bad Neustadt, Bad Neustadt an der Saale
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Städtisches Klinikum Dresden-Friedrichstadt, Dresden
  - Universitätsklinik an der Technischen Universität Dresden, Dresden
  - SRH Wald-Klinikum Gera GmbH, Gera
  - Universitätsklinikum Gießen und Marburg GmbH (UKGM), Giessen
  - Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Klinikum St. Georg gGmbH, Leipzig
  - Klinikum Leverkusen Service GmbH, Leverkusen
  - St.-Marien-Hospital GmbH, Lünen
  - Johannes Wesling Klinikum Minden, Minden
- Spain (3):
  - Hospital del Bierzo, León
  - Complejo Hospitalario de Ourense, Ourense
  - Hospital Universitario Marques de Valdecilla, Santander
- Switzerland (3):
  - CHUV - Centre Hospitalier Universitaire Vaudoise, Lausanne
  - Fondazione Cardiocentro Ticino, Lugano
  - Kantonsspital St. Gallen, Sankt Gallen

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 167 patients completed the informed consent process and signed the informed consent sheet. 166 patients successfully received the investigational device, the BM III.
Pre-assignment Details: March 18, 2020: temporary suspension of the enrollment due to the Covid-19 pandemic was announced. All investigators were informed about it and continuation of the follow-up phase. Instructions were given for the safety reporting, deviations from follow-up plan, and reporting of deviation in case these processes are impaired by Covid-19 situation. The suspension was lifted site by site based on pre-specified criteria between June 24, 2020 and February 5, 2021.
Groups:
- All Patients: BIOMONITOR III and BIOMONITOR IIIm: - Insertion of BIOMONITOR III or BIOMONITOR IIIm
  * three scheduled in-office follow-ups
  * 48-hour Holter ECG
Period: Overall Study
Arm/Group | All Patients
Started | 167
Completed | 116
Not Completed | 51
Not completed — Death | 3
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1
Not completed — Patient unable or unwilling to attend required visits | 8
Not completed — Drop-out according to protocol | 34

BASELINE CHARACTERISTICS:
Arm/Group | All Patients
Number analyzed (Participants) | 167
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67
  Male | 100
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Australia | 22
  Austria | 23
  Switzerland | 8
  Denmark | 3
  Spain | 14
  Germany | 97

OUTCOME MEASURES:

1. Primary Outcome: SADE-free Rate Until the 3-month Follow-up
Description: SADE-free rate related to BIOMONITOR III and BIOMONITOR IIIm including incision and insertion tool set until 3-month follow-up
Time Frame: 3 months
Population: All patients who either had a primary endpoint or who had reached 3 months of follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | All Patients
Number analyzed (Participants) | 159
Participants | 141
Statistical Analysis 1: Comparison: All Patients; The primary hypothesis evaluates the SADE free rate (pSADE_free) at 3 months. Ho: SADE-free rate through 3 months post-implant ≤ 90.0% Ha: SADE-free rate through 3 months post-implant > 90.0%; Test type: Other — single arm design; p = 0.05, t-test, 2 sided; SADE-free rate = 0.97, 95% CI 2-sided [0.9 to 1]

2. Secondary Outcome: R-wave Amplitude
Description: The secondary endpoint 1 evaluates the R-wave amplitude at the 1st follow-up and at 3-month follow-up by measuring both, the lowest and the highest amplitude value via the programmer.
Time Frame: 10 days to 4 weeks after insertion; 3-months
Reporting Status: Not Posted

3. Secondary Outcome: Noise Burden
Description: The secondary endpoint 2 evaluates the noise burden at the 1st follow-up and at 3-month follow-up by retrieving the percentage of noise via the programmer.
Time Frame: 10 days to 4 weeks after insertion; 3-months
Reporting Status: Not Posted

4. Secondary Outcome: Assessment of P-wave Visibility
Description: The secondary endpoint 3 evaluates the P-wave visibility at 1st, 3- and 12-month follow-up. The investigator will evaluate whether P-waves can be recognized in the stored sECGs showing sinus rhythm. The number of heart cycles and observed P-waves which can undoubtly be identified in ECGs will be assessed by the investigator.
Time Frame: 10 days to 4 weeks after insertion; 3-months
Reporting Status: Not Posted

5. Secondary Outcome: SADE-free Rate Until the 12-month Follow-up
Description: The secondary endpoint 4 is the SADE-free rate related to the BIOMONITOR III and BIOMONITOR IIIm 12 months after insertion.
Time Frame: 12-months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | All Patients
All-Cause Mortality (participants affected / at risk) | 3/167
Serious Adverse Events (participants affected / at risk) | 103/167
Other Adverse Events (participants affected / at risk) | 59/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=167)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Adverse drug reaction (General disorders) | 6 (6)
Antisynthetase syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 1 (1)
Aphasia (Nervous system disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 23 (24)
Atrial flutter (Cardiac disorders) | 3 (3)
Atrioventricular block (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 7 (7)
Blepharospasm (Eye disorders) | 1 (1)
Blood glucose increased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 7 (7)
Cardiac arrest (Cardiac disorders) | 8 (8)
Cardiac failure (Cardiac disorders) | 2 (2)
Cardiac tamponade (Cardiac disorders) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Chest pain (General disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Circulatory collapse (Vascular disorders) | 2 (2)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Condition aggravated (General disorders) | 2 (2)
Cor pulmonale (Cardiac disorders) | 1 (1)
Corona virus infection (Infections and infestations) | 2 (2)
Coronary artery disease (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 2 (2)
Cyst (General disorders) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device dislocation (Product Issues) | 2 (2)
Device extrusion (Product Issues) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Dilatation atrial (Cardiac disorders) | 1 (1)
Diverticulum (Gastrointestinal disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ejection fraction decreased (Investigations) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Heart rate increased (Investigations) | 1 (1)
Hiatus hernia (Gastrointestinal disorders) | 1 (1)
Hypertensive heart disease (Cardiac disorders) | 1 (1)
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Implant site haematoma (General disorders) | 1 (2)
Implant site haemorrhage (General disorders) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1)
Implant site pain (General disorders) | 2 (2)
Influenza (Infections and infestations) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 2 (2)
Lead dislodgement (Product Issues) | 1 (1)
Left atrial dilatation (Cardiac disorders) | 1 (1)
Left ventricular dysfunction (Cardiac disorders) | 1 (1)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 3 (4)
Nasal cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Oxygen saturation decreased (Investigations) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Respiratory tract infection (Infections and infestations) | 1 (1)
Right ventricular dilatation (Cardiac disorders) | 1 (1)
Scar pain (Skin and subcutaneous tissue disorders) | 1 (1)
Sinoatrial block (Cardiac disorders) | 1 (1)
Sinus arrest (Cardiac disorders) | 5 (5)
Sinus arrhythmia (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 4 (4)
Skin laceration (Injury, poisoning and procedural complications) | 1 (1)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 4 (5)
Syncope (Nervous system disorders) | 6 (6)
Tension headache (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 1 (1)
Tricuspid valve incompetence (Cardiac disorders) | 1 (1)
Troponin increased (Investigations) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Varices oesophageal (Gastrointestinal disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 5 (5)
Vertebral artery occlusion (Nervous system disorders) | 1 (1)
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Visual impairment (Eye disorders) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients (N=167)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Adverse drug reaction (General disorders) | 6 (6)
Amnesia (Nervous system disorders) | 1 (1)
Antisynthetase syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Anxiety disorder (Psychiatric disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Balance disorder (Nervous system disorders) | 1 (1)
Blood potassium decreased (Investigations) | 1 (1)
Bradycardia (Cardiac disorders) | 2 (2)
Cardiac arrest (Cardiac disorders) | 1 (1)
Chest discomfort (General disorders) | 2 (2)
Chest pain (General disorders) | 4 (5)
Chronic gastritis (Gastrointestinal disorders) | 1 (1)
Condition aggravated (General disorders) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Deafness (Ear and labyrinth disorders) | 1 (1)
Device dislocation (Product Issues) | 1 (1)
Device physical property issue (Product Issues) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Epilepsy (Nervous system disorders) | 1 (1)
Eye haemorrhage (Eye disorders) | 1 (1)
Facial bones fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 3 (5)
Fatigue (General disorders) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Heart rate increased (Investigations) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Implant site bruising (General disorders) | 2 (2)
Implant site haematoma (General disorders) | 3 (3)
Implant site haemorrhage (General disorders) | 2 (2)
Implant site infection (Infections and infestations) | 1 (1)
Implant site pain (General disorders) | 1 (1)
Implant site reaction (General disorders) | 1 (1)
Influenza like illness (General disorders) | 1 (1)
Intercepted medication error (Injury, poisoning and procedural complications) | 1 (1)
International normalised ratio fluctuation (Investigations) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Loss of consciousness (Nervous system disorders) | 1 (1)
Malaise (General disorders) | 2 (2)
Medical device site discomfort (General disorders) | 1 (1)
Munchausen's syndrome (Psychiatric disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthostatic intolerance (Nervous system disorders) | 1 (1)
Oversensing (Product Issues) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Patient dissatisfaction with device (Social circumstances) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Post procedural complication (Injury, poisoning and procedural complications) | 1 (1)
Pyoderma gangrenosum (Skin and subcutaneous tissue disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 2 (2)
Social problem (Social circumstances) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 3 (3)
Syncope (Nervous system disorders) | 3 (4)
Tachycardia (Cardiac disorders) | 1 (1)
Undersensing (Product Issues) | 2 (2)
Varicose vein (Vascular disorders) | 1 (1)
Ventricular extrasystoles (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 2 (2)
Visual impairment (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/10/NCT04025710/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-15): https://cdn.clinicaltrials.gov/large-docs/10/NCT04025710/SAP_001.pdf